CLINICAL TRIAL: NCT00588250
Title: Prospective Randomized Clinical Trial of Novel Implantation Promoting Medium (EmbryoGlue) to Improve IVF Success Rates
Brief Title: Clinical Trial of Novel Implantation Promoting Medium (EmbryoGlue) to Improve IVF Success Rates
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Implantation rate significantly lower in treatment group than Controls.
Sponsor: Mayo Clinic (Other)
Responsible Party: Dean E. Morbeck, PhD, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 876-04
Record Dates: First submitted 2007-12-22; First posted 2008-01-08 (Estimated); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Embryo Implantation; Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Other: EmbryoGlue
- B (No Intervention)

INTERVENTIONS:
Other: EmbryoGlue — G2 culture media from Vitrolife which contains hyaluronic acid
  Arms: A

SUMMARY:
Hypothesis: a special solution for improving human embryo implantation, when added to the solution during embryo transfer, will improve implantation rates in embryo transfers using previously frozen embryos.

DETAILED DESCRIPTION:
EmbryoGlue (TM) is added to embryo transfer solutions immediately prior to the transfer of frozen-thawed human embryos before placement of embryos into the patient uterus.

ELIGIBILITY:
Inclusion Criteria:

* Frozen embryo transfer patients, men over the age of 18 and women between the ages of 18 and 42 completed years (if using their own eggs and with embryos frozen before 39 completed years) or 18 to 50 completed years if using donated eggs.

Exclusion Criteria:

* Prior participation in this study, blastocyst transfers, single embryo transfer for medical reasons, prior embryo transfer with large amount of blood on the outside of the catheter, > or = 3 consecutive failed embryo transfers at Mayo Clinic (fresh or frozen-thawed cycles).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2003-05; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Pregnancy Rate | one month

SECONDARY OUTCOMES:
Implantation rate | two months

CONTACTS AND LOCATIONS:
Overall Officials: Dean E Morbeck, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States